CLINICAL TRIAL: NCT02000830
Title: A Four-Year Blinded Outcomes Follow-up Study of Patients Who Received Stannsoporfin or Placebo in Clinical Trial 64,185-204
Brief Title: Follow up Study of Patients Having Participated in Clinical Trial 64,185-204
Acronym: JASMINE_205
Status: Completed | Type: Observational
Sponsor: InfaCare Pharmaceuticals Corporation, a Mallinckrodt Company (Industry)
Responsible Party: Sponsor
Organization: Mallinckrodt (Industry)
Other Study IDs: 64,185-205
Record Dates: First submitted 2013-06-28; First posted 2013-12-04 (Estimated); Last update posted 2021-02-02 (Actual); Status verified 2021-01

CONDITIONS: Hyperbilirubinemia, Neonatal
Keywords: stannsoporfin
MeSH Terms: conditions — Hyperbilirubinemia, Neonatal | interventions — tin mesoporphyrin

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Prospective
Oversight: Data Monitoring Committee: No

GROUPS / COHORTS (3):
- Placebo: Participants received placebo during the earlier study
  Interventions: Drug: Placebo
- Stannsoporfin 3.0 mg/kg: Participants received Stannsoporfin 3.0 mg/kg during the earlier study
  Interventions: Drug: Stannsoporfin
- Stannsoporfin 4.5 mg/kg: Participants received Stannsoporfin 4.5 mg/kg during the earlier study
  Interventions: Drug: Stannsoporfin

INTERVENTIONS:
Drug: Stannsoporfin — Stannsoporfin administered by intramuscular (IM) injection
  Other Names: Experimental product
  Groups: Stannsoporfin 3.0 mg/kg; Stannsoporfin 4.5 mg/kg
Drug: Placebo — Matching placebo administered by IM injection
  Other Names: Matching Placebo
  Groups: Placebo

SUMMARY:
The objectives of this follow up study are to evaluate the long-term effects of stannsoporfin (Stanate) on the health, growth, and development of patients who received a single dose of stannsoporfin with PT used to treat hyperbilirubinemia compared with patients in the control (placebo plus PT) group in clinical trial 64,185-204.

DETAILED DESCRIPTION:
Outcomes will be based on the following variables:

Reported AEs and SAEs Hearing assessments Developmental assessments

ELIGIBILITY:
Inclusion Criteria:

* Patients who received IMP (stannsoporfin or placebo) in clinical trial 64,185-204
* Parents or guardians have given written informed consent to participate

Ages: 30 Days to 52 Months | Sex: All | Healthy Volunteers: No
Age Groups: Child
Study Population: Patients who received a single dose of trial medication in clinical trial 64,185-204.
Sampling Method: Probability Sample
Enrollment: 68 (Actual)
Dates: Start 2013-10-17 (Actual); Primary Completion 2020-02-28 (Actual); Study Completion 2020-02-28 (Actual)

PRIMARY OUTCOMES:
Reported adverse events (AEs) | 48-52 month

SECONDARY OUTCOMES:
Hearing assessments | 48 - 52 month
  Conventional audiometry will be performed by a qualified specialist. Any findings from a failed conventional audiology examination will be recorded
Developmental assessments | 48 - 52 month
  The Mullen Scales of Early Learning examination has been selected for its standardized measurement of developmental skills in multiple domains (gross motor, visual reception, fine motor, expressive language, and receptive language). Testing will be done at visits 1 and 2 by a healthcare individual trained to administer the test. The Mullen raw scores, T-scores, and age equivalents will be recorded.

CONTACTS AND LOCATIONS:
Overall Officials: Global Clinical Leader, MD, Study Chair — InfaCare Pharmaceuticals Corporation, a Mallinckrodt Company

IPD SHARING:
Plan to Share IPD: No